CLINICAL TRIAL: NCT05118490
Title: A Randomized Trial Comparing Treatment Completion of Daily Rifapentine & Isoniazid for One Month (1HP) To Weekly Rifapentine & Isoniazid For 3 Months (3HP) In Persons Living With HIV and in HIV-negative Household Contacts of Recently Diagnosed Tuberculosis Patients, The "One To Three" Trial
Brief Title: Comparing Treatment Completion Of Daily Rifapentine & Isoniazid For One Month (1HP) To Weekly High Dose Rifapentine & Isoniazid For 3 Months (3HP) In Persons Living With HIV and in Household Contacts of Recently Diagnosed Tuberculosis Patients
Acronym: 1 to 3
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Aurum Institute NPC (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00298999
Record Dates: First submitted 2021-10-26; First posted 2021-11-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: HIV Seropositivity; Tuberculosis; Household Contact
Keywords: Tuberculosis preventive treatment; rifapentine; HIV uninfected
MeSH Terms: conditions — HIV Seropositivity; Tuberculosis | interventions — Isoniazid

STUDY DESIGN:
Intervention Model Description: A randomization list will be generated prior to starting enrolment using random block sizes that are stratified by HIV status & country.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: People living with HIV infection without active TB (Experimental)
  Interventions: Drug: Daily rifapentine and isoniazid for 4 weeks; Drug: Weekly rifapentine and isoniazid for 12 weeks
- Group 2: HIV-negative household contacts of adults with rifampicin-sensitive pulmonary TB (Experimental)
  Interventions: Drug: Daily rifapentine and isoniazid for 4 weeks; Drug: Weekly rifapentine and isoniazid for 12 weeks

INTERVENTIONS:
Drug: Daily rifapentine and isoniazid for 4 weeks — Arm A: isoniazid (300mg) and rifapentine (600mg) daily for 4 weeks (1HP)
Drug: Weekly rifapentine and isoniazid for 12 weeks — Arm B: isoniazid (900mg) and rifapentine (900mg) weekly for 12 weeks (3HP)

SUMMARY:
A multicenter, randomized, stratified, open-label, phase IV trial among HIV-positive persons (PLHIV) on antiretroviral therapy (ART), or HIV-negative household contacts of patients with rifampicin-sensitive pulmonary tuberculosis (TB), who do not have evidence of active TB.

DETAILED DESCRIPTION:
Participants will be stratified by indication for tuberculosis (TB) preventive treatment (TPT) - HIV seropositive persons or HIV-negative household contact of person with infectious TB - and will receive either one of two TB preventive therapy regimens:

Group 1: People living with HIV infection without active TB

Arm A: isoniazid (300mg) and rifapentine (600mg) daily for 4 weeks (1HP)

Arm B: isoniazid (900mg) and rifapentine (900mg) weekly for 12 weeks (3HP)

Arm A (n=250): 250 participants age ≥13 years of age who are HIV seropositive and taking ART who do not have evidence of active TB will be recruited from local clinics. After being consented, screened, and randomized, participants in Arm A will receive the 1HP regimen once daily for 4 weeks (28 doses).

Study events include a health history, physical exam, TB symptom screen, symptom screen for adverse events (AEs), adherence checks during 1HP, and clinic visits at months 1, 2, and 6, at the least. Safety labs for liver function will be checked as clinically indicated.

Arm B (n=250): 250 participants age ≥13 years of age who are HIV seropositive and taking ART who do not have evidence of active TB will be recruited from local clinics. After being consented, screened, and randomized, participants in Arm B will receive the 3HP regimen once weekly for 12 weeks (12 doses).

Study events include a health history, physical exam, TB symptom screen, symptom screen for adverse events (AEs), adherence checks during 3HP, and clinic visits at months 1, 2, 3, and 6, at the least. Safety labs for liver function will be checked as clinically indicated.

Group 2: HIV-negative household contacts of newly diagnosed adults with rifampicin-sensitive pulmonary TB.

Arm A: isoniazid (300mg) and rifapentine (600mg) daily for 4 weeks (1HP)

Arm B: isoniazid (900mg) and rifapentine (900mg) weekly for 12 weeks (3HP)

Arm A (n=250): 250 participants age ≥13 years of age who are HIV-negative household contacts of adults with rifampicin-sensitive pulmonary TB who do not have evidence of active TB will be recruited from local clinics and households of active cases. After being consented, screened, and randomized, participants in Arm A will receive the 1HP regimen once daily for 4 weeks (28 doses).

Study events include a health history, physical exam, TB symptom screen, symptom screen for adverse events (AEs), adherence checks during 1HP, and clinic visits at months 1, 2, and 6, at the least. Safety labs for liver function will be checked as clinically indicated.

Arm B (n=250): 250 participants age ≥13 years of age who are HIV-negative household contacts of adults with rifampicin-sensitive pulmonary TB who do not have evidence of active TB will be recruited from local clinics and households of active cases. After being consented, screened, and randomized, participants in Arm B will receive the 3HP regimen once weekly for 12 weeks (12 doses).

Study events include a health history, physical exam, TB symptom screen, symptom screen for adverse events (AEs), adherence checks during 3HP, and clinic visits at months 1, 2, 3, and 6, at the least. Safety labs for liver function will be checked as clinically indicated.

ELIGIBILITY:
Group 1: HIV-positive adolescents and adults in South Africa and India

Inclusion criteria:

1. Age ≥ 13 years
2. Weight > 30 kg
3. HIV-seropositive
4. HIV viral load <400 copies/mL, defined as "virally suppressed," on an EFV or DTG-based ART regimen (see Section 3.6.2)
5. Candidates must meet WHO criteria for receiving TPT

Exclusion criteria:

1. Confirmed or suspected TB disease (evidenced by symptoms and/or clinical exam findings and/or chest radiographic findings suggestive of TB, positive mycobacterial culture or molecular TB testing or currently on TB treatment for active TB disease)
2. Likely to move from the study area during the study period
3. Known recent exposure to a TB case with resistance to isoniazid or rifampicin.
4. Previous treatment for active or latent TB for more than 30 days within the past 2 years
5. On nevirapine, etravirine, rilpivirine, PI-based, or raltegravir-containing ART regimens
6. Known sensitivity or intolerance to isoniazid or rifamycins
7. Suspected acute hepatitis or known chronic or unstable liver disease^
8. ALT > 3 times the upper limit of normal (ULN)
9. Total bilirubin > 2.5 times the ULN
10. Pregnancy or breastfeeding Females of childbearing potential who are unable or unwilling to use two forms of contraception**
11. On prohibited medications (see Appendix I)

Group 2: HIV-negative household contacts of an adult with confirmed pulmonary TB in Mozambique and Indonesia

Inclusion criteria:

1. Age ≥ 13 years
2. Weight > 30 kg
3. HIV-negative
4. Household contact of an adult with confirmed rifampicin-sensitive pulmonary TB
5. Candidates must meet WHO criteria for receiving TPT

Exclusion criteria:

1. Confirmed or suspected TB disease (evidenced by symptoms and/or clinical exam findings and/or chest radiographic findings suggestive of TB, positive mycobacterial culture or molecular TB testing or currently on TB treatment for active TB disease)
2. Likely to move from the study area during the study period
3. Known exposure to TB cases with resistance to isoniazid or rifampicin in the source case
4. Previous treatment for active or latent TB for >30 days within the past 2 years
5. Known sensitivity or intolerance to isoniazid or rifamycins
6. Suspected acute hepatitis or known chronic or unstable liver disease^
7. ALT > 3 times the upper limit of normal (ULN)
8. Total bilirubin > 2.5 times the ULN
9. Pregnancy or breastfeeding Females of childbearing potential who are unable or unwilling to use two forms of contraception**
10. On prohibited medications

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment adherence- self-report | from study entry at Week 0 through up to 8 weeks of 1HP (Group 1) or up to 24 weeks of 3HP (Group 2) , to be reported at end of trial
  Completion of TPT with >90% adherence documented by self-report (both groups, Arms A and B)
Treatment adherence- pill count | from study entry at Week 0 through up to 8 weeks of 1HP (Group 1) or up to 24 weeks of 3HP (Group 2) , to be reported at end of trial
  Completion of TPT with >90% adherence documented by pill count (both groups, Arms A and B)
Treatment adherence- electronic monitoring device (EMD) | from study entry at Week 0 through up to 8 weeks of 1HP (Group 1) or up to 24 weeks of 3HP (Group 2) , to be reported at end of trial
  Completion of TPT with >90% adherence documented by pill count (both groups, Arms A and B)
Adverse Events | from study entry at Day 0 through Month 6 (Week 24), to be reported at end of trial
  Occurrence of Grade 2 or higher targeted safety events (both groups, Arms A and B). Targeted safety events are hypersensitivity syndrome, rash, seizure, peripheral neuropathy, hepatotoxicity, nausea and vomiting, and drug-related fever.
Early treatment discontinuation | from study entry at Week 0 through up to 8 weeks of 1HP (Group 1) or up to 24 weeks of 3HP (Group 2), to be reported at end of trial
  discontinuation of study medications because of side effects (both groups, Arms A and B)

SECONDARY OUTCOMES:
Cost-effectiveness | from study entry at Week 0 through up to 8 weeks of 1HP (Group 1) or up to 24 weeks of 3HP (Group 2) , to be reported at end of trial
  Incremental cost-effectiveness of 1HP and 3HP (compared to each other, ^ months of isoniazid (6H), and no treatment) using a societal perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Churchyard, Study Chair — Aurum Institute
Locations (4):
- The Byramjee Jeejeebhoy Medical Centre (BJGMC-JHU) CRS, Pune, Maharashtra, India
- Yayasan KNCV - The Persahabatan Hospital, Jakarta, Jakarta, Jaya, Indonesia
- Fundação Aurum (The Aurum Institute Mozambique), Chokwé, Gaza Province, Mozambique
- The Aurum Institute: Gavin J Churchyard Legacy Centre, Klerksdorp, North West, South Africa

IPD SHARING:
Plan to Share IPD: No